CLINICAL TRIAL: NCT00137501
Title: Study of Different Doses of Nifedipine to Treat Preterm Labor
Brief Title: Two Dose Regimens of Nifedipine for the Management of Preterm Labor
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated because of difficulties in recruitement.
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Anwar Nassar, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: OGY.AN.01
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Labor, Premature
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): High dose Nifedpine arm
  Interventions: Drug: Nifedipine
- B (Other): Low dose Nifedipine arm
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — Arm A:
  Nifedipine 20 mg sublingual, repeated after 30 minutes if contractions do not decrease in intensity. Maintenance of 120-160 mgs of slow-release nifedipine daily for 48 hours.Once contractions cease, nifedipine will be maintained at 80-120 mg daily in divided doses up to 36 weeks.
  Arm B:
  Nifedipine 10 mg sublingual crushed, then 10 mg in 15 min, followed by 10 mg PO Q 15 mins PRN to a maximum of 40 mg in the first hour. Maintenance of 60-80 mgs of slow-release nifedipine daily for 48 hours. Once contractions cease, nifedipine will be maintained at 60 mg daily in divided doses up to 36 weeks.
  Other Names: Adalat, Nifedicor

SUMMARY:
Preterm birth is one of the most important causes of perinatal morbidity and mortality worldwide. Prevention and treatment of preterm labor is important, not as an end in itself, but as a means of reducing adverse events for the neonate. A wide range of tocolytics, drugs used to suppress uterine contractions, have been tried. Magnesium sulfate (MgSO4) is the most widely used tocolytic at the American University of Beirut Medical Center despite the fact that an effective tocolytic role of MgSO4 has never been established. Moreover, the currently available data are suggestive of deleterious fetal effects of MgSO4 in the setting of preterm labor to the extent that some authorities are recommending abandoning it for routine use as a tocolytic therapy. Calcium channel blockers have the ability to inhibit contractility in smooth muscle cells. Consequently, nifedipine has emerged as an effective and rather safe alternative tocolytic agent for the management of preterm labor after several studies have shown that the use of nifedipine in comparison with other tocolytics is associated with a more frequent successful prolongation of pregnancy, resulting in significantly fewer admissions of newborns to the neonatal intensive care unit, and is associated with a lower incidence of respiratory distress syndrome. The unequivocal impact of this method of tocolysis on short term postponement of delivery and the opportunity that this provides for affecting in-utero transfer and steroid administration has prompted many investigators to recommend focusing future trials on testing different dose regimens of nifedipine. To the best of the investigators' knowledge, no study comparing two different dose regimens of nifedipine has been previously published in the literature. The objective of their study is to compare the effectiveness of a high versus a low dose regimen in a total of 200 patients admitted with the diagnosis of preterm labor between 24 and 34 weeks of gestation. In addition, the investigators' study will try to assess the safety profile of the 2 dose regimens on the mother and the neonate by assessing a selected number of outcome variables. The data generated will be used to change their protocol for managing patients presenting with threatened preterm delivery and will fill the existing gap regarding the most effective and safest dose regimen of nifedipine in such patients.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

Inclusion criteria:

* All pregnant women diagnosed with preterm labor defined as regular contractions associated with cervical change between 24 and 34 weeks of gestation.

Exclusion criteria:

* Multiple pregnancy
* Preterm rupture of membranes
* Congenital fetal malformations
* IUGR (intra uterine growth restriction)
* Previous tocolysis this pregnancy
* Chorioamnionitis
* Cervical dilation > 4 cms
* Maternal medical conditions such as renal insufficiency, hepatic insufficiency, or myasthenia gravis
* Non-reassuring fetal heart rate
* Maternal hypotension, defined as a blood pressure < 90/50 mm Hg

Randomization procedure:

Randomization envelopes will be prepared by means of a random number table. After informed consent is obtained, the next numbered opaque envelope will be opened to assign each patient to receive either the low or high nifedipine dose regimen. Because of the different doses of nifedipine, neither patients nor physicians will be blinded to treatment allocation.

Routine studies and procedures:

* A baseline ECG will be performed before starting the medication.
* All patients will receive a 500-mL intravenous bolus of isotonic sodium chloride solution unless they have clinical volume overload, followed by a maintenance administration of 125 mL/h.
* Maternal blood pressure and heart rate will be recorded every 15 minutes as long as the patient is in labor and every 4 hours thereafter.
* Fetal heart rate and uterine activity were monitored continuously throughout the study period.
* All patients eligible for the study will receive antibiotic prophylaxis for Group B Streptococcal infection (IV Pen G or Ampicillin) for at least 48 hours, pending the vaginorectal swab culture that is done routinely on every patient presenting with preterm labor.
* All patients will receive one course of 12 mg betamethasone intramuscularly every 24 hours for 48 hours to promote fetal lung maturation and a rescue dose if they present in labor again at < 34 weeks of gestation.

Interventions:

First arm (high dose):

Nifedipine (Adalat®) 20 mg sublingual crushed, repeated after 30 minutes if contractions do not decrease in intensity. Maintenance of 120-160 mgs of slow-release nifedipine (Nifedicor®) daily for 48 hours (30 mg Q 6 hrs up to a maximum of 40 mg Q 6 hrs). Once contractions cease, nifedipine will be maintained at 80-120 mg daily in divided doses up to 36 weeks of gestation on an outside basis.

Second arm (low dose):

Nifedipine (Adalat®) 10 mg sublingual crushed, then 10 mg sublingual in 15 min, followed by 10 mg PO Q 15 mins PRN to a maximum of 40 mg in the first hour. Maintenance of 60-80 mgs of slow-release nifedipine (Nifedicor®) daily for 48 hours (20 mg Q 8 hrs or 20 mg Q 6 hrs). Once contractions cease, nifedipine will be maintained at 60 mg daily in divided doses up to 36 weeks of gestation.

* Tocolysis will be considered to be achieved when uterine activity decrease to <4 contractions/h with the absence of cervical change.
* If patients continue to have uterine activity after 6 hours or have cervical dilatation >2 cm after admission examination, they could be switched to another tocolytic regimen, namely intravenous MgSO4 or intravenous ritodrine.

Written Consent:

The written consent will be handed to every pregnant patient eligible for this study. She will be given enough time to read it and decide whether she is willing to participate in the trial.

Outcome variables studied:

* Speed of onset of uterine quiescence
* Uterine quiescence at 6 hours of initiating therapy
* Delivery >48 hours from initiation of therapy
* Delivery >7 days from initiation of therapy
* Delivery <37 weeks of gestation
* Delivery at <34 weeks of gestation
* Side effects to nifedipine
* Maternal adverse drug reactions requiring cessation of treatment
* Antepartum hemorrhage
* Maternal length of hospital stay
* Pregnancy prolongation
* Postpartum hemorrhage
* Birthweight
* Apgar score <7 at 5 min
* Admission to NICU
* Mechanical ventilation
* RDS (respiratory distress syndrome)
* IVH all grades
* Neonatal nursery stay
* Neonatal jaundice
* NEC (Necrotizing enterocolitis)
* Neonatal death

Side effects associated with nifedipine include a mild decrease in blood pressure and a rise in pulse, headache, flushing, dizziness and nausea.

Data Collection:

The initial information in the data sheets will be filled by the resident in charge of delivery suite. However, the follow up on the response of the patients to the medication and data regarding the maternal side effects and neonatal outcome will be filled by a part time research assistant.

Statistical Analysis:

Statistical analysis will be performed using the SPSS statistical package. Categoric data like maternal characteristics, the rates of neonatal morbidity and mortality will be compared using Chi square when sample sizes support the approximation. Otherwise, categorical data will be analyzed with two-tailed Fisher exact test if the expected cell frequencies were small. Continuous variables will be compared by Student t test if assumptions of normality and homogeneity of variances appeared to be reasonable. Unpaired variables and differences in distributions will be compared using the Mann-Whitney test. Neonatal outcomes will be analyzed comparing the total number of affected neonates in each group. A p-value <0.05 will be considered statistically significant.

Proposed budget:

Personnel:

A part time research assistant with "BS" background 450,000 L.L./ month x 29 months =13,050,000 L.L.

Tasks expected:

Completing the data sheets:

* F/U on response of mother to tocolysis and assessing maternal side effects
* F/U on the neonates and getting information about the neonatal outcome variables
* Data entry

Medical supplies:

Medications will be provided through the pharmacy.

Compensation for patients:

None.

The total amount of money needed in Lebanese pounds:

13,050,000 L.L./year.

Time frame:

* May 2003 - May 2006 - Collection of data and randomization of patients to the 2 arms of the study
* June 2006 - Sep 2006 - Follow up on patients that were randomized during the first 5 months of 2006 to get information about their pregnancy outcome
* Oct 2006 - Nov 2006 - Data analysis and writing the final paper

Data collection will be under the direct supervision of the principal investigator.

Percent of time spent by principal investigator on this proposal: 20% of research time which accounts for about 20% of time allocated for research activities.

Co-Investigators' Role:

* Dr Usta will help in data analysis and in writing the final paper (5% of research time)
* Dr Mroueh will help in writing the final paper (5% of research time). Two Investigational Drug forms will be used since this trial will involve the same drug nifedipine in 2 different forms Adalat® and Nifedicor®.

Principal Investigator:

Anwar Nassar, MD, Assistant Professor, American University of Beirut Medical Center, Department of Obstetrics and Gynecology

Co-Investigators:

Ihab Usta, MD, Associate Professor, American University of Beirut Medical Center, Department of Obstetrics and Gynecology

Adnan Mroueh, MD, Professor, American University of Beirut Medical Center, Department of Obstetrics and Gynecology

REFERENCES:

Assessment of Risk Factors for Preterm Birth. ACOG practice bulletin, Number 31, October 2001.

Mittendorf R, Dambrosia J, Pryde PG, Lee KS, Gianopoulos JG, Besinger RE, Tomich PG. Association between the use of antenatal magnesium sulfate in preterm labor and adverse health outcomes in infants. Am J Obstet Gynecol;186(6):1111-8. June 2002.

Gyetvai K, Hannah ME, Hodnett ED, Ohlsson A. Tocolytics for preterm labor: a systematic review. Obstet Gynecol;94(5 Pt 2):869-77. Nov 1999.

Mittendorf R, Covert R, Elin R, Pryde PG, Khoshnood B, Lee KS. Umbilical cord serum ionized magnesium level and total pediatric mortality. Obstet Gynecol; 98(1):75-8. July 2001.

Weerakul W, Chittacharoen A, Suthutvoravut S. Nifedipine versus terbutaline in management of preterm labor. Int J Gynaecol Obstet;76(3):311-3. Mar 2002.

Papatsonis DN, Van Geijn HP, Ader HJ, Lange FM, Bleker OP, Dekker GA. Nifedipine and ritodrine in the management of preterm labor: a randomized multicenter trial. Obstet Gynecol;90(2):230-4. Aug 1997.

Larmon JE, Ross BS, May WL, Dickerson GA, Fischer RG, Morrison JC. Oral nicardipine versus intravenous magnesium sulfate for the treatment of preterm labor. Am J Obstet Gynecol;181(6):1432-7. Dec1999.

Koks CA, Brolmann HA, de Kleine MJ, Manger PA. A randomized comparison of nifedipine and ritodrine for suppression of preterm labor. Eur J Obstet Gynecol Reprod Biol;77(2):171-6. Apr 1998.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women diagnosed with preterm labor defined as regular contractions associated with cervical change between 24 and 34 weeks of gestation

Exclusion Criteria:

* Multiple pregnancy
* Preterm rupture of membranes
* Congenital fetal malformations
* IUGR (intra uterine growth restriction)
* Previous tocolysis in this pregnancy
* Chorioamnionitis
* Cervical dilation > 4 cms
* Maternal medical conditions such as renal insufficiency, hepatic insufficiency, or myasthenia gravis
* Non-reassuring fetal heart rate
* Maternal hypotension, defined as a blood pressure < 90/50 mmHg

Ages: 17 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2003-05; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Uterine quiescence at 48 hours of initiation of tocolysis | 2 days

SECONDARY OUTCOMES:
Speed of uterine quiescence, remaining undelivered at >48 hours and >7 days after tocolysis, delivery <34 and 37 weeks of gestation, hours to quiescence, gestational age, maternal drug reactions, hospital stay, neonatal morbidities &neonatal death. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anwar H Nassar, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon